CLINICAL TRIAL: NCT02547025
Title: Personalized Treatment for Refractory H Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS13-CT12-17
Record Dates: First submitted 2015-09-08; First posted 2015-09-11 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; third-line therapy; antibiotic susceptibility; Eradication
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Clarithromycin; Tetracycline; Levofloxacin; bismuth tripotassium dicitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rabeprazole+3 antibiotics (Experimental): patients who have positive result of culture with equal to or more than three susceptible antibiotics are treated by non-bismuth quadruple therapy (rabeprazole 20 mg q.d.s. and three effective antibiotics) for 14 days
  Interventions: Drug: rabeprazole+3 antibiotics
- rabeprazole+bismuth+2 antibiotics (Experimental): patients who have positive result of culture with one or two susceptible antibiotics are treated by bismuth-containing therapy (rabeprazole 20 mg q.d.s., bismuth subcitrate 120 mg q.d.s. and all the effective antibiotics) for 14 days
  Interventions: Drug: rabeprazole+bismuth+2 antibiotics
- rabeprazole+amox+tetr+levo (Active Comparator): patients who have negative result of culture or whose culture data are unavailable will be treated by (rabeprazole 20 mg q.d.s, amoxicillin 500 mg q.d.s., tetracycline 500 mg q.d.s. and levofloxacin 500 mg o.d.) for 14 days
  Interventions: Drug: rabeprazole+amox+tetr+levo

INTERVENTIONS:
Drug: rabeprazole+3 antibiotics — (rabeprazole 20 mg q.d.s. and three effective antibiotics) for 14 days.
  Other Names: rabeprazole 20 mg; amoxicillin 1g; clarithromycin 500mg; metrondazole 250mg; tetracycline 500mg; levofloxacin 500mg
  Arms: rabeprazole+3 antibiotics
Drug: rabeprazole+bismuth+2 antibiotics — (rabeprazole 20 mg q.d.s., bismuth subcitrate 120 mg q.d.s. and all the effective antibiotics) for 14 days.
  Other Names: rabeprazole 20 mg; bismuth subcitrate 120 mg; amoxicillin 1g; clarithromycin 500mg; metrondazole 250mg; tetracycline 500mg; levofloxacin 500mg
  Arms: rabeprazole+bismuth+2 antibiotics
Drug: rabeprazole+amox+tetr+levo — (rabeprazole 20 mg q.d.s, amoxicillin 500 mg q.d.s., tetracycline 500 mg q.d.s. and levofloxacin 500 mg o.d.) for 14 days.
  Other Names: rabeprazole 20 mg; bismuth subcitrate 120 mg; tetracycline 500mg; levofloxacin 500mg
  Arms: rabeprazole+amox+tetr+levo

SUMMARY:
In this study, the investigators develop a personalized treatment according to culture-guided antibiotics plus high-dose proton-pump inhibitor and bismuth to treat refractory H pylori infection.

DETAILED DESCRIPTION:
They are categorized into three groups: (1) patients who have positive result of culture with equal to or more than three susceptible antibiotics are treated by non-bismuth quadruple therapy (rabeprazole 20 mg q.d.s. and three effective antibiotics), (2) patients who have positive result of culture with one or two susceptible antibiotics are treated by bismuth-containing therapy (rabeprazole 20 mg q.d.s., bismuth subcitrate 120 mg q.d.s. and all the effective antibiotics), and (3) patients who have negative result of culture or whose culture data are unavailable will be treated by (rabeprazole 20 mg q.d.s, amoxicillin 500 mg q.d.s., tetracycline 500 mg q.d.s. and levofloxacin 500 mg o.d.) for 14 days.

ELIGIBILITY:
Inclusion Criteria:

H pylori-infected adult patients with at least two previous failed eradication attempts will be enrolled in this study after giving informed consent.

* positive results of both rapid urease test and histology,
* a positive result of Urea breath test,
* or a positive result of culture

Exclusion Criteria:

* ingestion of antibiotics, bismuth, or proton-pump inhibitor within the prior 4 weeks,
* patients with allergic history to the medications used,
* patients with previous gastric surgery,
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia),
* pregnant women.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants in Which H. Pylori Was Eradicated | eight weeks after the end of anti-H pylori therapy
  To assess eradication efficacy,repeated endoscopy with rapid urease test, histological examination and culture or Urea breath test.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Current European concepts in the management of Helicobacter pylori infection. The Maastricht Consensus Report. European Helicobacter Pylori Study Group. Gut. 1997 Jul;41(1):8-13. doi: 10.1136/gut.41.1.8. PMID 9274464
- [Background] Megraud F. H pylori antibiotic resistance: prevalence, importance, and advances in testing. Gut. 2004 Sep;53(9):1374-84. doi: 10.1136/gut.2003.022111. No abstract available. PMID 15306603
- [Background] Luther J, Higgins PD, Schoenfeld PS, Moayyedi P, Vakil N, Chey WD. Empiric quadruple vs. triple therapy for primary treatment of Helicobacter pylori infection: Systematic review and meta-analysis of efficacy and tolerability. Am J Gastroenterol. 2010 Jan;105(1):65-73. doi: 10.1038/ajg.2009.508. Epub 2009 Sep 15. PMID 19755966
- [Background] De Francesco V, Margiotta M, Zullo A, Hassan C, Troiani L, Burattini O, Stella F, Di Leo A, Russo F, Marangi S, Monno R, Stoppino V, Morini S, Panella C, Ierardi E. Clarithromycin-resistant genotypes and eradication of Helicobacter pylori. Ann Intern Med. 2006 Jan 17;144(2):94-100. doi: 10.7326/0003-4819-144-2-200601170-00006. PMID 16418408
- [Background] Graham DY, Shiotani A. New concepts of resistance in the treatment of Helicobacter pylori infections. Nat Clin Pract Gastroenterol Hepatol. 2008 Jun;5(6):321-31. doi: 10.1038/ncpgasthep1138. Epub 2008 Apr 29. PMID 18446147
- [Background] Goodwin CS, Marshall BJ, Blincow ED, Wilson DH, Blackbourn S, Phillips M. Prevention of nitroimidazole resistance in Campylobacter pylori by coadministration of colloidal bismuth subcitrate: clinical and in vitro studies. J Clin Pathol. 1988 Feb;41(2):207-10. doi: 10.1136/jcp.41.2.207. PMID 3280609
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Wu DC, Hsu PI, Tseng HH, Tsay FW, Lai KH, Kuo CH, Wang SW, Chen A. Helicobacter pylori infection: a randomized, controlled study comparing 2 rescue therapies after failure of standard triple therapies. Medicine (Baltimore). 2011 May;90(3):180-185. doi: 10.1097/MD.0b013e31821c9d1c. PMID 21512411
- [Background] Gisbert JP. "Rescue" regimens after Helicobacter pylori treatment failure. World J Gastroenterol. 2008 Sep 21;14(35):5385-402. doi: 10.3748/wjg.14.5385. PMID 18803350
- [Background] Hojo M, Miwa H, Nagahara A, Sato N. Pooled analysis on the efficacy of the second-line treatment regimens for Helicobacter pylori infection. Scand J Gastroenterol. 2001 Jul;36(7):690-700. doi: 10.1080/003655201300191941. PMID 11444467
- [Background] Lee BH, Kim N, Hwang TJ, Lee SH, Park YS, Hwang JH, Kim JW, Jeong SH, Lee DH, Jung HC, Song IS. Bismuth-containing quadruple therapy as second-line treatment for Helicobacter pylori infection: effect of treatment duration and antibiotic resistance on the eradication rate in Korea. Helicobacter. 2010 Feb;15(1):38-45. doi: 10.1111/j.1523-5378.2009.00735.x. PMID 20302588
- [Background] Kuo CH, Hu HM, Kuo FC, Hsu PI, Chen A, Yu FJ, Tsai PY, Wu IC, Wang SW, Li CJ, Weng BC, Chang LL, Jan CM, Wang WM, Wu DC. Efficacy of levofloxacin-based rescue therapy for Helicobacter pylori infection after standard triple therapy: a randomized controlled trial. J Antimicrob Chemother. 2009 May;63(5):1017-24. doi: 10.1093/jac/dkp034. Epub 2009 Feb 26. PMID 19246508
- [Background] Saad RJ, Schoenfeld P, Kim HM, Chey WD. Levofloxacin-based triple therapy versus bismuth-based quadruple therapy for persistent Helicobacter pylori infection: a meta-analysis. Am J Gastroenterol. 2006 Mar;101(3):488-96. doi: 10.1111/j.1572-0241.2006.00637.x. PMID 16542284
- [Background] Wong WM, Gu Q, Chu KM, Yee YK, Fung FM, Tong TS, Chan AO, Lai KC, Chan CK, Wong BC. Lansoprazole, levofloxacin and amoxicillin triple therapy vs. quadruple therapy as second-line treatment of resistant Helicobacter pylori infection. Aliment Pharmacol Ther. 2006 Feb 1;23(3):421-7. doi: 10.1111/j.1365-2036.2006.02764.x. PMID 16423001
- [Background] Cammarota G, Martino A, Pirozzi G, Cianci R, Branca G, Nista EC, Cazzato A, Cannizzaro O, Miele L, Grieco A, Gasbarrini A, Gasbarrini G. High efficacy of 1-week doxycycline- and amoxicillin-based quadruple regimen in a culture-guided, third-line treatment approach for Helicobacter pylori infection. Aliment Pharmacol Ther. 2004 Apr 1;19(7):789-95. doi: 10.1111/j.1365-2036.2004.01910.x. PMID 15043520
- [Background] Savarino V, Zentilin P, Pivari M, Bisso G, Raffaella Mele M, Bilardi C, Borro P, Dulbecco P, Tessieri L, Mansi C, Borgonovo G, De Salvo L, Vigneri S. The impact of antibiotic resistance on the efficacy of three 7-day regimens against Helicobacter pylori. Aliment Pharmacol Ther. 2000 Jul;14(7):893-900. doi: 10.1046/j.1365-2036.2000.00780.x. PMID 10886045
- [Background] Megraud F, Lamouliatte H. Review article: the treatment of refractory Helicobacter pylori infection. Aliment Pharmacol Ther. 2003 Jun 1;17(11):1333-43. doi: 10.1046/j.1365-2036.2003.01592.x. PMID 12786627
- [Background] Megraud F. Adjuvant therapy for Helicobacter pylori eradication: role of lansoprazole shown in vitro. J Clin Gastroenterol. 1995;20 Suppl 1:S24-7. PMID 7673610
- [Background] Padol S, Yuan Y, Thabane M, Padol IT, Hunt RH. The effect of CYP2C19 polymorphisms on H. pylori eradication rate in dual and triple first-line PPI therapies: a meta-analysis. Am J Gastroenterol. 2006 Jul;101(7):1467-75. doi: 10.1111/j.1572-0241.2006.00717.x. PMID 16863547
- [Background] Schwab M, Schaeffeler E, Klotz U, Treiber G. CYP2C19 polymorphism is a major predictor of treatment failure in white patients by use of lansoprazole-based quadruple therapy for eradication of Helicobacter pylori. Clin Pharmacol Ther. 2004 Sep;76(3):201-9. doi: 10.1016/j.clpt.2004.05.002. PMID 15371981
- [Background] Furuta T, Sugimoto M, Kodaira C, Nishino M, Yamade M, Uotani T, Ikuma M, Shirai N. The dual therapy with 4 times daily dosing of rabeprazole and amoxicillin as the 3rd rescue regimen for eradication of H. pylori. Hepatogastroenterology. 2010 Sep-Oct;57(102-103):1314-9. PMID 21410079
- [Background] Hsu PI, Lai KH, Tseng HH, Lo GH, Lo CC, Lin CK, Cheng JS, Chan HH, Ku MK, Peng NJ, Chien EJ, Chen W, Hsu PN. Eradication of Helicobacter pylori prevents ulcer development in patients with ulcer-like functional dyspepsia. Aliment Pharmacol Ther. 2001 Feb;15(2):195-201. doi: 10.1046/j.1365-2036.2001.00903.x. PMID 11148437
- [Background] Hsu PI, Lai KH, Tseng HH, Liu YC, Yen MY, Lin CK, Lo GH, Huang RL, Huang JS, Cheng JS, Huang WK, Ger LP, Chen W, Hsu PN. Correlation of serum immunoglobulin G Helicobacter pylori antibody titers with histologic and endoscopic findings in patients with dyspepsia. J Clin Gastroenterol. 1997 Dec;25(4):587-91. doi: 10.1097/00004836-199712000-00007. PMID 9451668
- [Background] Hsu PI, Lai KH, Chien EJ, Lin CK, Lo GH, Jou HS, Cheng JS, Chan HH, Hsu JH, Ger LP, Hsu PN, Tseng HH. Impact of bacterial eradication on the cell proliferation and p53 protein accumulation in Helicobacter pylori-associated gastritis. Anticancer Res. 2000 Mar-Apr;20(2B):1221-8. PMID 10810425
- [Background] Peng NJ, Lai KH, Liu RS, Lee SC, Tsay DG, Lo CC, Tseng HH, Huang WK, Lo GH, Hsu PI. Endoscopic 13C-urea breath test for the diagnosis of Helicobacter pylori infection. Dig Liver Dis. 2003 Feb;35(2):73-7. doi: 10.1016/s1590-8658(03)00014-8. PMID 12747623
- [Background] Peng NJ, Lai KH, Liu RS, Lee SC, Tsay DG, Lo CC, Tseng HH, Huang WK, Lo GH, Hsu PI. Clinical significance of oral urease in diagnosis of Helicobacter pylori infection by [13C]urea breath test. Dig Dis Sci. 2001 Aug;46(8):1772-8. doi: 10.1023/a:1010626225949. PMID 11508681
- [Background] Kita T, Sakaeda T, Aoyama N, Sakai T, Kawahara Y, Kasuga M, Okumura K. Optimal dose of omeprazole for CYP2C19 extensive metabolizers in anti-Helicobacter pylori therapy: pharmacokinetic considerations. Biol Pharm Bull. 2002 Jul;25(7):923-7. doi: 10.1248/bpb.25.923. PMID 12132671